CLINICAL TRIAL: NCT03616808
Title: The Influence of Thromboelastometry-identified Haemostatic Changes on Haemorrhagic Progression of Intracranial Injury and Clinical Outcome in Patients With Isolated Traumatic Brain Injury
Brief Title: Thromboelastometry-identified Haemostatic Changes in Isolated Traumatic Brain Injury
Acronym: THROMBIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, MARIUS RIMAITIS, PhD student, Lithuanian University of Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V2
Record Dates: First submitted 2018-07-13; First posted 2018-08-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Coagulation Disorder; Brain Injuries, Traumatic; Bleeding
Keywords: Traumatic brain injury; Craniotomy; Goal-directed treatment; Thromboelastometry
MeSH Terms: conditions — Hemostatic Disorders; Brain Injuries, Traumatic; Hemorrhage

STUDY DESIGN:
Intervention Model Description: A case-control study. Conventional management patients are considered as "controls" whereas goal-directed management patients will be considered "cases".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional therapy (No Intervention): Intraoperative haemostatic treatment is based on conventional coagulation assays.
- Goal-directed therapy (Active Comparator): Thromboelastometry-guided haemostatic treatment is provided intraoperatively.
  Interventions: Other: Thromboelastometry-guided haemostatic treatment

INTERVENTIONS:
Other: Thromboelastometry-guided haemostatic treatment — Administration of blood products and/or procoagulants is based on thromboelastometric assays.
  Arms: Goal-directed therapy

SUMMARY:
A prospective open-label case-control study will be performed aiming to assess the utility of thromboelastometry (ROTEM) for identification of hemostatic changes, goal-directed coagulation management, and prognosis of intracranial hemorrhagic injury progression as well as clinical outcome in patients with isolated traumatic brain injury. Patients undergoing craniotomy to treat traumatic brain injury will be enrolled. All patients will undergo standard perioperative coagulation analysis (APTT, PT, INR, fibrinogen levels, platelet count), whereas ROTEM-guided group will additionally be tested with ROTEM. "Cases" will be managed according to a ROTEM-based algorithm, and "Controls" will be treated as usual (based on clinical judging). Comparative analysis of acquired demographic, clinical and laboratory data will be performed. The investigators believe that ROTEM results could provide better insight into perioperative coagulation changes, be beneficial to patient blood management, and result in better outcome.

DETAILED DESCRIPTION:
Aim of the study:

To assess the utility of thromboelastometry for identification of hemostatic changes, goal-directed coagulation management, and prognosis of intracranial hemorrhagic injury progression as well as clinical outcome in patients with isolated traumatic brain injury.

Objectives:

To evaluate perioperative prevalence and characteristics of thromboelastometry identified coagulopathy in neurosurgical patients with isolated traumatic brain injury; To assess the correlation between routine laboratory test results and thromboelastometric findings; To evaluate the influence of thromboelastometric findings and goal-directed coagulation management on the progression of intracranial hemorrhagic injury; To evaluate the utility of thromboelastometry for goal-directed coagulation management, and its possible influence on clinical outcome.

Study background:

Traumatic brain injury still accounts for a considerable proportion of preventable deaths worldwide. The prevalence of coagulation derangements among patients with traumatic brain injury (TBI) is high and approximates 30 % (1,2). The main hypothesis explaining the development of coagulopathy in the absence of massive bleeding is extensive release of tissue factor from the damaged brain tissue and subsequent over-activation of coagulation leading to consumption of coagulation substrates. The presence of coagulopathy in the setting of TBI is associated with high risk of intracranial hemorrhagic insult progression and death (3,4). Many authors investigating coagulopathy associated with traumatic brain injury have used routine coagulation tests, such as APTT, PT, INR, fibrinogen levels. However, those tests do not reflect the overall clot quality and reflect only separate parts of the coagulation process.

Craniotomy for traumatic brain injury is an urgent high-risk procedure presenting a serious challenge for the anesthesiology team. Significant, diffuse bleeding is not infrequent, and the spectrum of neurosurgical hemostatic options is limited. Moreover, even small amounts of intracranial blood may be life-threatening. Therefore the maintenance of optimal physiologic clotting capacity is crucial. Literature data investigating the use of ROTEM in TBI patients is still limited (5,6).

The investigators believe that thromboelastometry could provide novel insights into the dynamic coagulation changes of TBI patients. Moreover, it could serve as a clinical tool for targeted coagulation management in the perioperative period of patients undergoing craniotomies for intracranial traumatic hematomas, and prove beneficial for patient outcome.

Materials and methods:

A prospective open-label case-control study will be performed. Adult isolated traumatic brain injury patients undergoing craniotomy and will be enrolled. Required sample size was calculated based on the average number of craniotomies performed to treat traumatic brain injury during the past five years in a tertiary neurosurgical centre. The investigators plan to enroll 70 patients into the ROTEM-guided group (Cases), and 70 patients into the conventional therapy group (Controls). All patients will undergo standard coagulation analysis (APTT, PT, INR, fibrinogen levels, platelet count) preoperatively, and 3 days postoperatively, whereas ROTEM-guided group patients will additionally be tested with ROTEM (EXTEM, INTEM, FIBTEM, APTEM). Coagulation management decisions in the ROTEM-guided group will be made according to a ROTEM-based algorithm for goal-directed hemostatic therapy. Conventional therapy group will be treated as usual. Perioperative demographic, clinical and laboratory data of study patients will be registered. Early neurological state (on postoperative days 1,2,3,7, and until discharge) will be assessed according to the Glasgow coma scale. Late neurological outcome (6 and 12 months postoperatively) will be assessed according to Glasgow outcome scale. Comparative analysis of Case and Control groups will be performed. Perioperative prevalence and characteristics of coagulopathy in neurosurgical patients with isolated traumatic brain injury will be estimated. Correlation between routine laboratory test results and thromboelastometric findings will be assessed. The influence of thromboelastometric findings and goal-directed coagulation management on the progression of intracranial hemorrhagic injury will be assessed. The influence of goal-directed coagulation management on clinical outcome will be evaluated.

Anticipated scientific and clinical benefits:

The investigators believe that ROTEM results could provide better insight into perioperative coagulation changes, be beneficial to patient blood management, and result in better outcome.

ELIGIBILITY:
Inclusion Criteria:

* Isolated traumatic brain injury (within 48 hours) (AIS head >= 3)
* Urgent craniotomy is necessary
* A written informed consent is acquired from the patient or his/her representative

Exclusion Criteria:

* Refusal / inability to acquire an informed consent
* Significant trauma to other body regions (AIS other regions >= 3)
* Data on significant chronic hepatic or hematologic illness
* Use of oral anticoagulants or antiplatelet agents
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Mortality of patients in both groups
Early neurological state according to Glasgow coma scale | 30 days
  Glasgow coma scale (GCS) is used to objectively assess the level of consciousness after neurological injury according to best eye (range 1 to 4), verbal (range 1 to 5) and motor (range 1 to 6) response of the patient. Eye, verbal and motor scores are summed to give the total Glasgow coma score (range 3 to 15). The lowest possible GCS (the sum) is 3 (deep coma or death), while the highest is 15 (fully awake person).

SECONDARY OUTCOMES:
Coagulation abnormalities on conventional coagulation assays and ROTEM | 72 hours
  The number of patients with abnormal results of PT (prothrombin time), INR (international normalized ratio), APTT (activated partial thromboplastin time), fibrinogen concentration, platelet count and/or any abnormal thromboelastometric (ROTEM) parameter
Progressive hemorrhagic injury | 30 days
  Evidence of new or increased intracranial hemorrhagic injury
Clinical outcome according to Glasgow outcome score | Up to 1 year
  The Glasgow Outcome Score (GOS) is used to divide patients with traumatic brain injury into groups (range 1 to 5) that allow standardised descriptions of the objective degree of recovery as follows:
  1. Death
  2. Persistent vegetative state - Severe damage with prolonged state of unresponsiveness and a lack of higher mental functions
  3. Severe disability - Severe injury with permanent need for help with daily living
  4. Moderate disability - No need for assistance in everyday life, employment is possible but may require special equipment
  5. Low disability - Light damage with minor neurological and psychological deficits

OTHER OUTCOMES:
Correlation between conventional coagulation assays and ROTEM parameters | 72 hours
  The number of cases with corresponding results (both abnormal (or normal) conventional coagulation assays and ROTEM parameters) vs. the number of cases with conflicting results (abnormal (or normal) conventional coagulation assays, but normal (or abnormal) ROTEM parameters); Correlation between PT and EXTEM CT (thromboelastometric measure of clotting time in the extrinsic coagulation pathway); Correlation between APTT and INTEM CT (thromboelastometric measure of clotting time in the intrinsic coagulation pathway); Correlation between fibrinogen concentration and FIBTEM MCF (thromboelastometric measure of maximum clot firmness in the fibrinogen polymerisation assay); Correlation between platelet count and EXTEM MCF (thromboelastometric measure of maximum clot firmness in the extrinsic coagulation pathway); Correlation between platelet count and INTEM MCF (thromboelastometric measure of maximum clot firmness in the intrinsic coagulation pathway)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wafaisade A, Lefering R, Tjardes T, Wutzler S, Simanski C, Paffrath T, Fischer P, Bouillon B, Maegele M; Trauma Registry of DGU. Acute coagulopathy in isolated blunt traumatic brain injury. Neurocrit Care. 2010 Apr;12(2):211-9. doi: 10.1007/s12028-009-9281-1. PMID 19806475
- [Background] Harhangi BS, Kompanje EJ, Leebeek FW, Maas AI. Coagulation disorders after traumatic brain injury. Acta Neurochir (Wien). 2008 Feb;150(2):165-75; discussion 175. doi: 10.1007/s00701-007-1475-8. Epub 2008 Jan 2. PMID 18166989
- [Background] Maegele M. Coagulopathy after traumatic brain injury: incidence, pathogenesis, and treatment options. Transfusion. 2013 Jan;53 Suppl 1:28S-37S. doi: 10.1111/trf.12033. PMID 23301970
- [Background] de Oliveira Manoel AL, Neto AC, Veigas PV, Rizoli S. Traumatic brain injury associated coagulopathy. Neurocrit Care. 2015 Feb;22(1):34-44. doi: 10.1007/s12028-014-0026-4. PMID 25052157
- [Background] Brazinova A, Majdan M, Leitgeb J, Trimmel H, Mauritz W; Austrian Working Group on Improvement of Early TBI Care. Factors that may improve outcomes of early traumatic brain injury care: prospective multicenter study in Austria. Scand J Trauma Resusc Emerg Med. 2015 Jul 16;23:53. doi: 10.1186/s13049-015-0133-z. PMID 26179747
- [Background] Schochl H, Solomon C, Traintinger S, Nienaber U, Tacacs-Tolnai A, Windhofer C, Bahrami S, Voelckel W. Thromboelastometric (ROTEM) findings in patients suffering from isolated severe traumatic brain injury. J Neurotrauma. 2011 Oct;28(10):2033-41. doi: 10.1089/neu.2010.1744. Epub 2011 Sep 23. PMID 21942848
- [Derived] Rimaitis M, Cechanoviciute V, Bilskiene D, Balciuniene N, Vilcinis R, Rimaitis K, Macas A. Dynamic Changes of Hemostasis in Patients with Traumatic Brain Injury Undergoing Craniotomy: Association with in-Hospital Mortality. Neurocrit Care. 2023 Jun;38(3):714-725. doi: 10.1007/s12028-022-01639-4. Epub 2022 Dec 5. PMID 36471184